CLINICAL TRIAL: NCT04644510
Title: Feasability of Lung Ultrasonography in General Practice: A Multicentic, Observational and Descriptive Study
Brief Title: Feasability of Lung Ultrasonography in General Practice
Acronym: AmBulUs
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-023; 2019-A00205-52 (Other: ID-RCB)
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Ultrasonography; Education; General Practice
Keywords: Ultrasonography; General Practice; Feasability; Lung ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung ultrasonography group: Patient which benefited from a Lung ultrasonography during the medical consultation
  Interventions: Device: Lung ultrasonography

INTERVENTIONS:
Device: Lung ultrasonography — Standardized eight-point Lung ultrasonography

SUMMARY:
A major barrier to ultrasonography in general practice (GP) is the time restriction of their medical consultation. We aimed to evaluate the feasibility of lung ultrasonography (LUS) realized by general practitioners (GP's) into their medical consultation.

A prospective, observational, multi-centric and open study conducted in 3 different centers by 15 GP in France. Patient receiving LUS were recruited from December 2019 to January 2020. GP's were all novices and received a training course by LUS expert before the study. Eight-points LUS exam was recorded, timed, and interpreted by GP's.

Among the 111 LUS performed, 110 LUS were interpreted. Time duration was 4 (3-5) min with 13% of LUS superior to 5 minutes. There was no significant difference in time duration after stratification by age. Patients were mainly satisfied after receiving LUS, and 80% of patients had a better understanding about their disease due to US realization.

In this first prospective, and multicenter study, involving patients consulting in General Practice, we found that LUS seems to be feasible by GP's in a medical consultation. We showed that LUS can be performed fast enough for a GP consultation, and easy to learn. These findings will need to be valided in a randomized and controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 3 months; lung ultrasonography performed by GP

Exclusion Criteria:

* Age < 3 months or rejection to participate to the study

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients consulting their family physician
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Duration of Lung Ultrasonography | 2 months

SECONDARY OUTCOMES:
Time limit exceeded lung ultrasonography | 2 months
  Superior to 5 minutes
Interpretation of lung ultrasonography images | 2 months
Stratification by age | 2 months
  3 groups : < 18 years-old, 18-65 years-old, > 65 years-old
Survey results | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No